CLINICAL TRIAL: NCT01160653
Title: Cognitive and Motor Training After Stroke for Everyday Walking Restoration
Brief Title: Cognitive & Motor Training After Stroke For Everyday Walking Restoration
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Never funded
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UNF1
Record Dates: First submitted 2010-04-26; First posted 2010-07-12 (Estimated); Last update posted 2014-02-25 (Estimated); Status verified 2014-02

CONDITIONS: Stroke
Keywords: stroke; Gait training; Cognitive Training
MeSH Terms: conditions — Stroke | interventions — Cognitive Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Gait training and Cognitive Training
  Interventions: Device: FES-IM; Other: Cognitive training
- 2 (No Intervention): Able Bodied

INTERVENTIONS:
Device: FES-IM — implantable Functional Electrical Stimulation
  Arms: 1
Other: Cognitive training — training of impaired cognitive processes
  Arms: 1

SUMMARY:
The purpose of this study is to test a unique, combined cognitive and motor intervention designed to restore safe, more normal coordinated gait components into the real world environment for individuals with stroke.

ELIGIBILITY:
Inclusion Criteria:

* greater than or equal to 6 months post stroke
* ability to give informed consent
* impaired gait
* medically stable

Exclusion Criteria:

* pacemaker
* unstable/uncontrolled medical condition(s)

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-08; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Coordinated Components of gait using the Gait Assessment and Intervention Tool (G.A.I.T.) | post treatment

CONTACTS AND LOCATIONS:
Overall Officials: Janis Daly, PhD MS, Principal Investigator — VA Medical Center-Cleveland
Locations (1):
- VA Medical Center, Cleveland, Cleveland, Ohio, United States